CLINICAL TRIAL: NCT03209609
Title: A Multi-center, Randomized, Within-subject-controlled, Open Label Study of the Safety and Effectiveness of VEST, Venous External Support
Brief Title: VEST Venous Graft External Support Pivotal Study
Acronym: VEST Pivotal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Graft Solutions Ltd. (Industry)
Collaborators: International Center for Health Outcomes and Innovation Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CD0131
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery bypass
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: In each patient, one SVG bypass will be randomized to be supported by the VEST, while another will not be supported and serve as control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- VEST supported vein graft (Experimental): Coronary artery bypass vein graft supported with the VEST implant
  Interventions: Device: VEST; Procedure: Coronary artery bypass vein grafts
- Standard of care vein grafts (Active Comparator): Coronary artery bypass vein grafts
  Interventions: Procedure: Coronary artery bypass vein grafts

INTERVENTIONS:
Device: VEST — External support for vein grafts, cobalt chrome braid
  Arms: VEST supported vein graft
Procedure: Coronary artery bypass vein grafts — Bypass coronary arteries with autologous saphenous vein grafts

SUMMARY:
Prospective, multi-center, randomized, within-subject-controlled , trial, enrolling patients with multi vessel atherosclerotic coronary artery disease, scheduled to undergo SVG CABG with arterial grafting of IMA to LAD and two or more saphenous vein grafts. In each patient, one SVG bypass will be randomized to be supported by the VEST, while another will not be supported and serve as control. Thus, the full cohort will provide a basis for comparison between two sets of SVGs: A VEST supported set; and an unsupported set.

DETAILED DESCRIPTION:
Clinical significance:

Coronary artery bypass grafting (CABG) remains the gold standard treatment for patients with multi-vessel coronary artery disease. Despite the proposed benefits of multiple arterial grafts, autologous saphenous vein grafts (SVGs) are still the most frequently used bypass conduits in CABG. Progressive SVG failure after CABG remains a key limitation to the long-term success of surgery.

Objective:

Coronary artery bypass grafting (CABG) remains the gold standard treatment for patients with multi-vessel coronary artery disease. Despite the proposed benefits of multiple arterial grafts, autologous saphenous vein grafts (SVGs) are still the most frequently used bypass conduits in CABG. Progressive SVG failure after CABG remains a key limitation to the long-term success of surgery.

Study design:

Prospective, multi-center, randomized, within-subject-controlled , trial, enrolling patients with multi vessel atherosclerotic coronary artery disease, scheduled to undergo SVG CABG with arterial grafting of IMA to LAD and two or more saphenous vein grafts. In each patient, one SVG bypass will be randomized to be supported by the VEST, while another will not be supported and serve as control. Thus, the full cohort will provide a basis for comparison between two sets of SVGs: A VEST supported set; and an unsupported set.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, inclusive of release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documentation.
2. Age 21 years or older.
3. Planned and scheduled on-pump CABG.
4. Two or more vein grafts to native vessels having at least 75% stenosis and comparable runoff.
5. IMA graft indicated for the LAD. Additional arterial grafts may be considered based on practice guidelines.
6. Appropriately sized and accessible target coronary arteries, with a minimum diameter of 1.5 mm and adequate vascular bed (without significant distal stenosis), as assessed by pre-operative cardiac angiography and verified by diameter gauging intraoperatively.

Exclusion Criteria:

1. Concomitant non-CABG cardiac surgical procedure.
2. Prior cardiac surgery.
3. Emergency CABG surgery.
4. Contraindication for on-pump CABG with cardioplegic arrest (e.g. severely calcified aorta).
5. Calcification at the intended anastomotic sites, as assessed upon opening of the chest and before randomization.
6. Severe vein varicosity as assessed after vein harvesting and before randomization.
7. History of clinical stroke within 3 months prior to randomization.
8. Severe renal dysfunction (Cr>2.0 mg/dL).
9. Documented or suspected untreated diffuse peripheral vascular disease such as: carotid stenosis or claudication of the extremities.
10. Concomitant life-threatening disease likely to limit life expectancy to less than two years.
11. Inability to tolerate or comply with required guideline-based post-operative drug regimen (antiplatelet plus statin) and/or inability to take aspirin.
12. Inability to comply with required follow-ups including angiographic imaging methods (e.g. contrast allergy).
13. Concurrent participation in an interventional (drug or device) trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Intimal hyperplasia area/graft occlusion | 1 year
  Intimal hyperplasia (plaque+media) area [mm2] as assessed by IVUS at 12 months. Occluded vessels are accounted for in the analysis of the primary endpoint

SECONDARY OUTCOMES:
Lumen diameter uniformity | 1 year
  Lumen diameter uniformity, assessed by angiography for each graft separately and expressed by the Fitzgibbon classification (22), on a 3-point ordinal scale
vein graft failure | 1 year
  Graft Failure (≥50% stenosis) by cardiac angiography

OTHER OUTCOMES:
MACCE | annually over 5 years
  Major adverse cardiac and cerebrovascular events

CONTACTS AND LOCATIONS:
Overall Officials: John Puskas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Daniel Goldstein, MD, Principal Investigator — Montefiore Medical Center
Locations (17):
- United States (14):
  - University of Southern California, Los Angeles, California
  - Lutheran Hospital of Indiana, Fort Wayne, Indiana
  - University of Maryland Baltimore, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Mount Sinai St Luke's, New York, New York
  - New York Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Scott & White Research Institute, The Heart Hospital Baylor Plano, Plano, Texas
  - University of Virginia, Charlottesville, Virginia
- Canada (3):
  - London Health Sciences Centre, University Hospital, London, Ontario
  - Institut de Cardiologie de Montréal, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldstein DJ, Puskas JD, Alexander JH, Chang HL, Gammie JS, Marks ME, Iribarne A, Vengrenyuk Y, Raymond S, Taylor BS, Yarden O, Orion E, Dagenais F, Ailawadi G, Chu MWA, DiMaio JM, Narula J, Moquete EG, O'Sullivan K, Williams JB Jr, Crestanello JA, Jessup M, Rose EA, Scavo V, Acker MA, Gillinov M, Mack MJ, Gelijns AC, O'Gara PT, Moskowitz AJ, Bagiella E, Voisine P. External Support for Saphenous Vein Grafts in Coronary Artery Bypass Surgery: A Randomized Clinical Trial. JAMA Cardiol. 2022 Aug 1;7(8):808-816. doi: 10.1001/jamacardio.2022.1437. PMID 35675092